CLINICAL TRIAL: NCT06866002
Title: Study of Diabetes' Risk Factors and Accelerated Aging According to Socio-economic Status in a Population From the North of France - 3-year Follow-up
Acronym: PrévenDIAB 2
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Coralie BERTHIER, Research prevention center manager, Institut Pasteur de Lille
Other Study IDs: 2024-A02836-41
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Prediabetes
Keywords: Risk factors; Precarious; Accelerated aging; (Pre) diabetes
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Glucose Intolerance | interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Main Group: observational descriptive cohort
  Interventions: Other: Biological analysis, Physical examination and Questionnaires
- Sub group: Case control study
  Interventions: Other: Physical examination and Questionnaires

INTERVENTIONS:
Other: Biological analysis, Physical examination and Questionnaires — Biological analysis, Physical examination and questionnaires will be performed for all patients of the main group.
  Groups: Main Group
Other: Physical examination and Questionnaires — In addition to exams for the main group, there will be 2 additional examinations (arterial stiffness) for the patients of the subgroup and others questionnaires.
  Groups: Sub group

SUMMARY:
Populations in precarious situations or with low socio-economic status are at greater risk of diabetes and accelerated ageing. Depending on the population studied, the factors that may explain these health inequalities are not unequivocal and remain poorly understood.

Northern France, which is particularly affected by socio-economic disparities, has one of the highest diabetes prevalence rates in mainland France. This is why the researchers wanted to study the clinical, biological, social and behavioral risk factors for the onset of diabetes and accelerated aging in a large population in northern France.

A 2021 study aimed to characterize the population (a majority of whom (55%) suffer from precarious conditions) who came to the Institut Pasteur de Lille for their health check-up, in order to study risk factors to better explain these health inequalities.

This research consisted of a descriptive observational cross-sectional study carried out on 2233 volunteers (main group) over 18 months, and a complementary analytical case-control study involving 216 participants (sub-group).

At present, we are planning a 3-year follow-up of the cohort. Participants will be recontacted for a new health check-up at the Centre d'examen de Santé de l'Institut Pasteur de Lille. At the end of the health check-up, participants will be interviewed by PrévenDIAB study investigators to collect the same data as initially collected, with the exception of some data we deemed unnecessary.

DETAILED DESCRIPTION:
Primary Objective : To measure changes in fasting glycemic control after 3 years in PrevenDIAB-1 study participants according to socioeconomic status

Primary efficacy endpoint : fasting plasma glucose and Hb1Ac

* Conversion rate of glycemic status (worsening, stable, improving) according to EPICES score
* Prevalence of pre-diabetes/diabetes (T0 and T 3 years) according to EPICES score

Secondary objectivesspecific to the main group :

* Observe the evolution of anthropometric factors such as BMI (weight), waist circumference and various measures of body composition, and determine their role in the evolution of glycemia.
* Observe the evolution of clinical, biological, metabolomic, behavioral and environmental factors, and determine their role in the evolution of glycemia.
* Measure the impact of PrevenDIAB-1 (+/- prevention intervention) on changes in behaviour and health perception according to socio-economic status (has the completion of a health check-up enabled people to resume a course of care and/or raise awareness/engage in prevention?)
* Gather information on subjects' possible participation in preventive actions, define them (type, duration, indication, etc.) and assess their potential impact on risk factors.
* Propose a personalized care pathway for different risk profiles (roadmap defined for people with diabetes or morbid obesity, for example), create a city-hospital link and follow up with subjects by telephone at 6 months to obtain their feedback/opinions on the management of their pathology.

Secondary Objectives specific to the sub-group:

* Measure changes in the following subgroup parameters:

  * physical activity
  * sleep
  * alcohol consumption
  * frailty
  * arterial stiffness
  * cognitive status
* Determine the link with pre-diabetes and diabetes.
* Obtain qualitative data by setting up focus groups on the co-creation of a "space of trust" promoting health empowerment.

  * This work will be carried out by a "health and human sciences" post-doc in 2025.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the PrévenDIAB study

Exclusion Criteria:

* Subject participating in another clinical study or in a period of exclusion from another study and incompatible with PrévenDIAB-2 follow-up
* Refusal to participate in study
* Scheduling impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Populations in precarious situations or with low socio-economic status are at greater risk of developing diabetes and of accelerated ageing. Depending on the populations studied, the factors that may explain these health inequalities are not unequivocal and remain poorly understood.
  The Hauts-de-France region, which is particularly affected by socio-economic disparities, has one of the highest prevalence rates of diabetes in mainland France. That's why we want to study the clinical, biological, social and behavioral risk factors for diabetes onset and accelerated aging in a large population in northern France.
  Our study aims to characterize the population of consultants at the Centre d'Examens de Santé l'Institut Pasteur de Lille, the majority of whom (55%) suffer from precarious conditions, in order to study the risk factors that may better explain these health inequalities.
  This population will be monitored every 3 years to assess changes in the various parameters.
Sampling Method: Non-Probability Sample
Enrollment: 2011 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose and Hb1Ac | Day 0
  Conversion rate of glycemic status (worsening, stable, improving) according to EPICES score. Prevalence of pre-diabetes/diabetes (T0 and T 3 years) according to EPICES score

SECONDARY OUTCOMES:
Prevalence ratio of (pre)diabetes calculated for clinical, biological and behavioral/environmental explanatory variables | Day 0
  In %
Prevalence ratio of (pre) diabetes and accelerated aging according to the socio-economic status | Day 0
  In %
Risk (odds Ratio) of (pre) diabetes and accelerated aging according to social, economic, cultural and professional status | Until Day 90
  Without units
Risk (odds Ratio) of (pre) diabetes and accelerated aging for assessed exposures | Until Day 90
  Without units

CONTACTS AND LOCATIONS:
Overall Officials: Philippe FROGUEL, Study Chair — PhD PRECIDIAB; Matthias VANDESQUILLE, Study Director — PhD PRECIDIAB
Locations (1):
- Institut Pasteur de Lille, Lille, Hauts de France, France

IPD SHARING:
Plan to Share IPD: No